CLINICAL TRIAL: NCT03325205
Title: MR Guided tDCS: The Effect of Repeated Transcranial Direct Current Stimulation on Cognitive Functioning in Alzheimer's Disease
Brief Title: MR Guided tDCS in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: Helse Nord (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/794 (REK)
Record Dates: First submitted 2017-09-04; First posted 2017-10-30 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Alzheimer's Disease
Keywords: Transcranial direct current stimulation; Neuromodulation; Individualizing brain stimulation; Neuropsychology
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Participants receive anodal tDCS over DLPFC. Each sessions lasts for 20 minutes, with a total of 15 stimulations: 6 acute sessions, 9 maintenance sessions.
  Interventions: Other: Anodal tDCS
- Sham tDCS (Sham Comparator): Participants receive sham tDCS over DLPFC. Each sessions lasts for 20 minutes, with a total of 15 stimulations: 6 acute sessions, 9 maintenance sessions.
  Interventions: Other: Sham tDCS

INTERVENTIONS:
Other: Anodal tDCS — Anodal Transcranial direct current stimulation (tDCS) is a non- invasive brain stimulation technique. Low intensity current (1-2 mA) is induced to increase excitability, stimulate plasticity and enhance cognitive functions.
  Arms: Active tDCS
Other: Sham tDCS — The electrodes are placed over the same areas as in the anodal tDCS condition. Participants will receive sham tDCS instead of anodal tDCS
  Arms: Sham tDCS

SUMMARY:
The purpose of the study is to investigate the effect of High Density- tDCS (HD- tDCS) on cognitive function in Alzheimer's Disease. One anode and four return electrodes are placed over DLPFC, where low intensity current (2mA) is induced to the surface of the scalp. Electrode placement is individualized for each participant. Participants will undergo 15 stimulations, with a duration of 20 minutes each. All patients will undergo neuropsychological assessment and MRI evaluation.

DETAILED DESCRIPTION:
The project will be run as a Randomized Controlled Trial (RCT), where patients will be randomized to receive either active anodal tDCS or sham tDCS. The performance on neuropsychological tests will be the primary outcome variables in the present project. In addition, whole brain MRI volume measures will be used to measure specific effects of tDCS treatment. Electrode placement is individualized for each participant with brain modeling techniques.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's Disease, mild and moderate stage

Exclusion Criteria:

* Other neurological diseases or injuries
* Stroke
* Cancer
* Psychiatric disorders (moderate/ severe depression, psychosis)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Performance on Neuropsychological tests | 4 months
  Compare scores before and after tDCS stimulation

SECONDARY OUTCOMES:
Hippocampal volume | 4 months
  Compare performance on neuropsychological tests to hippocampal volume. Here we are looking at correlations between hippocampal thickness, performance on neuropsychological tests and effect of tDCS.

CONTACTS AND LOCATIONS:
Overall Officials: Per M Aslaksen, Professor, Principal Investigator — University of Tromso
Locations (1):
- Department of Psychology, University of Northern Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rasmussen ID, Boayue NM, Mittner M, Bystad M, Gronli OK, Vangberg TR, Csifcsak G, Aslaksen PM. High-Definition Transcranial Direct Current Stimulation Improves Delayed Memory in Alzheimer's Disease Patients: A Pilot Study Using Computational Modeling to Optimize Electrode Position. J Alzheimers Dis. 2021;83(2):753-769. doi: 10.3233/JAD-210378. PMID 34366347